CLINICAL TRIAL: NCT01213589
Title: The VIRTUE Post Marketing Surveillance Registry - VALIANT Thoracic Stent Graft Evaluation For the Treatment of Descending Thoracic Aortic Dissections
Brief Title: The VIRTUE Post Marketing Surveillance Registry
Acronym: VIRTUE
Status: Completed | Type: Observational
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDTVIRTUE001
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-10

CONDITIONS: Aortic Dissection
Keywords: descending; thoracic; aortic; dissection; Valiant; Medtronic; Type B; VIRTUE; stent
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Descending thoracic aortic dissection: Patients diagnosed with a descending thoracic aortic dissection and who are amenable to stent-graft operation. The patient had an indication for treatment by either endovascular stent graft implantation for either an acute, sub-acute or chronic Type B dissection.

SUMMARY:
The purpose of this post-market release registry is to collect additional information concerning safety, performance and health economic data with respect to the Medtronic VALIANT Thoracic Stent Graft with the Xcelerant Delivery System in the treatment of descending thoracic aortic dissections.

DETAILED DESCRIPTION:
The patient device for use in this registry is the Medtronic VALIANT Thoracic Stent Graft System that received CE mark approval in March 2005.

The Medtronic VALIANT Thoracic Stent Graft with Xcelerant Delivery System is designed to treat diseases of the descending thoracic aorta including but not limited to aneurysms and dissections. The VALIANT Stent Graft is designed to exclude the aneurysm, the false lumen or site of rupture and restore the blood flow through the stent graft lumen. The device is intended for use either in patients who are candidates for conventional surgical repair, and in patients who are not candidates for conventional surgical repair due to pre-existing risk factors.

This registry is a prospective, non-randomized, single-arm, multi-center, European clinical registry with patients diagnosed with descending thoracic aortic dissection.

For this registry standard hospital procedures with respect to patient interventional care for thoracic aortic diseases will be followed.

This is a descriptive registry in which no specific hypotheses will be statistically tested.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be more than or equal to 18 years of age; or older if required by local regulations.
* Patient has an indication for treatment by either endovascular stent graft implantation for either an acute, sub-acute or chronic Type B dissection.
* Patient is amenable for stent-graft treatment (in accordance with the IFU).
* The patient is willing and able to cooperate with registry procedures and required follow-up visits.
* The patient or legal guardian has signed a patient informed consent form, including data privacy authorization (this criteria is not applicable for patients presenting in emergency with ruptured dissection and for whom legal representative is not available informed consent can be requested after surgical procedure).

Exclusion Criteria:

* Patients with a thoracic dissection for which optimal treatment is observation and medical management.
* Patient with current - non aortic - medical condition with a life expectancy less than one year.
* The patient is participating in another device or drug study (patient must have completed the follow-up phase of any previous study at least 30 days prior to enrolment in this registry).
* Time interval between medical indication for surgical intervention and endovascular procedure exceeds 4 months (122 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a descending thoracic aortic dissection and who are amenable to stent-graft operation will be enrolled in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Thompson, Prof., Principal Investigator — St George's Hospital; D. Gasparini, Dr., Principal Investigator — Azienda Ospedaliera "Santa Maria della Misericordia"; R. Fattori, Prof., Principal Investigator — Ospedale Sant'Orsola Malpighi; P. Cao, Dr., Principal Investigator — Unità di Chirurgia Vascolare, Ospedale R. Silvestrini; G. Garzón, Dr., Principal Investigator — Hospital Universitario La Paz; E. Ros, Prof., Principal Investigator — Hospital Clínico Universitario San Cecilio; B. Rylski, Dr., Principal Investigator — Universitätsklinikum Freiburg; S. Huptas, Dr., Principal Investigator — Universitätsklinikum Essen; I. Degrieck, Dr., Principal Investigator — Onze-Lieve-Vrouw Ziekenhuis; D. Dai-DoDo, Prof., Principal Investigator — Universitätsspital Bern, Inselspital; H. Roos, Dr., Principal Investigator — Sahlgrenska University Hospital; R. Heijmen, Dr., Principal Investigator — St. Antonius Hospital; N. Cheshire, Prof., Principal Investigator — St Mary's NHS Trust; C. Nienaber, Dr, Principal Investigator — University School of Medicine Rostock

REFERENCES:
- [Result] Virtue Registry Investigators. The VIRTUE Registry of type B thoracic dissections--study design and early results. Eur J Vasc Endovasc Surg. 2011 Feb;41(2):159-66. doi: 10.1016/j.ejvs.2010.08.016. Epub 2010 Oct 16. PMID 20952217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of study patients in the Registry began in the medical clinics on 5 December 2006 and was completed on 26 August 2009.
Pre-assignment Details: No subject got excluded after enrollment
Groups:
- Acute: Patients diagnosed with a descending thoracic aortic dissection and who are amenable to stent-graft operation. The patient had an indication for treatment by either endovascular stent graft implantation for an acute Type B dissection.
- Sub-acute: Patients diagnosed with a descending thoracic aortic dissection and who are amenable to stent-graft operation. The patient had an indication for treatment by either endovascular stent graft implantation for a sub-acute Type B dissection.
- Chronic: Patients diagnosed with a descending thoracic aortic dissection and who are amenable to stent-graft operation. The patient had an indication for treatment by either endovascular stent graft implantation for a chronic Type B dissection.
Period: Overall Study
Arm/Group | Acute | Sub-acute | Chronic
Started | 50 | 24 | 26
Completed | 37 | 19 | 18
Not Completed | 13 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute | Sub-acute | Chronic | Total
Number analyzed (Participants) | 50 | 24 | 26 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 18 | 19 | 62
  >=65 years | 25 | 6 | 7 | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (14.1) | 59.7 (11.0) | 58.8 (10.9) | 61.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 6 | 24
  Male | 38 | 18 | 20 | 76
Region of Enrollment [Number; unit: participants]
  Europe | 50 | 24 | 26 | 100

OUTCOME MEASURES:

1. Primary Outcome: Disease-, Procedure- or Device-related Mortality at 12 Months Post-procedure
Description: Disease, device or procedure-related mortality at 12 months post-procedure, defined as any death related to the device, to the disease or to the surgical procedure occurring in the period of 365 days following the day of the implant procedure.
Time Frame: 12 months post-procedure
Measure: Number; unit: participants
Arm/Group | Acute | Sub-acute | Chronic
Number analyzed (Participants) | 50 | 24 | 26
participants | 9 | 1 | 1

2. Secondary Outcome: Safety
Description: * All causes mortality
  * Disease-, procedure- or device-related mortality
Time Frame: 30 days or at discharge, 3/6/12/24/36 months
Measure: Number; unit: participants
Arm/Group | Acute | Sub-acute | Chronic
Number analyzed (Participants) | 50 | 24 | 26
participants | 9 | 1 | 6

3. Secondary Outcome: Efficacy/Performance
Description: - Technical Success Technical success, defined as a composite of (i) successful introduction and deployment of at least one Valiant Thoracic Stent Graft at the intended location, (ii) successful coverage of the proximal entry tear, (iii) no immediate conversion to open surgery during the same intervention, (iv) absence of death within 24 hours post-procedure, and (v) the absence of significant graft twist, kink or obstruction by intra-operative measurements
Time Frame: 30 days or at discharge, 3/6/12/24/36 months
Measure: Number; unit: participants
Arm/Group | Acute | Sub-acute | Chronic
Number analyzed (Participants) | 50 | 24 | 26
participants | 49 | 24 | 25

4. Secondary Outcome: Freedom of Re-intervention
Description: Kaplan-Meier estimate of freedom from secondary procedures by clinical group.
Time Frame: 30 days or at discharge, 3/6/12/24/36 months
Measure: Number; unit: Percentage Event Free
Arm/Group | Acute | Sub-acute | Chronic
Number analyzed (Participants) | 50 | 24 | 26
Percentage Event Free | 71.7 | 68.8 | 66.7

5. Secondary Outcome: Freedom From Disease-, Procedure- or Device-related Major Complications
Description: Complications were assigned a severity score (according SVS scores) so that degrees of morbidity can be assessed and compared. A moderate complication indicates the need for significant intervention, prolongation of hospitalization more than 24 hours, and at most, minor permanent disability that does not preclude normal daily activity. A severe complication necessitates major surgical or medical intervention, may be associated with prolonged convalescence, is usually accompanied by prolonged or permanent disability, and may result in death. Both moderate and severe complications are considered as major complications.
  Kaplan-Meier estimate of freedom from disease-, procedure-, or device-related major complications by clinical group.
Time Frame: through 36 months
Measure: Number; unit: Percentage Event Free
Arm/Group | Acute | Sub-acute | Chronic
Number analyzed (Participants) | 50 | 24 | 26
Percentage Event Free | 37.4 | 41.3 | 40.3

6. Secondary Outcome: Freedom From Disease-, Procedure-, or Device-related Severe Complications
Description: Complications were assigned a severity score (according SVS scores) so that degrees of morbidity can be assessed and compared. A severe complication necessitates major surgical or medical intervention, may be associated with prolonged convalescence, is usually accompanied by prolonged or permanent disability, and may result in death.
  Kaplan-Meier estimate of freedom from disease-, procedure-, or device-related severe complications
Time Frame: through 36 months
Measure: Number; unit: Percentage Event Free
Arm/Group | Acute | Sub-acute | Chronic
Number analyzed (Participants) | 50 | 24 | 26
Percentage Event Free | 67.8 | 75.0 | 64.1

7. Secondary Outcome: Clinical Success
Description: Clinical success was defined as: (i) successful introduction and deployment of the Valiant Thoracic Stent Graft at the intended location; (ii) successful coverage of the proximal entry tear; (iii) no immediate conversion to open surgery;(iv) absence of surgical open repair or endovascular re-intervention; (v) absence of death related to aortic disease or treatment; (vi) absence of graft thrombosis, obstructions, twists or kinks; (vii) absence of graft migration;(viii) absence of graft integrity failure; (ix) at the level of the ostium of the LSA, the more proximal entry tear of the dissection, the largest section of the thoracic aorta, and at the first image/slice available with upper part of the liver:
  Absence of true lumen decrease in diameter (≥ 5 mm is significant) Absence of increase in total aortic diameter (≥ 5 mm is significant)
Time Frame: through 36 months
Measure: Number; unit: participants
Arm/Group | Acute | Sub-acute | Chronic
Number analyzed (Participants) | 50 | 24 | 26
participants | 18 | 9 | 8

ADVERSE EVENTS:
Arm/Group | Acute | Sub-acute | Chronic
Serious Adverse Events (participants affected / at risk) | 35/50 | 15/24 | 19/26
Other Adverse Events (participants affected / at risk) | 3/50 | 2/24 | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acute (N=50) | Sub-acute (N=24) | Chronic (N=26)
Pulmonary Complications (General) (Respiratory, thoracic and mediastinal disorders) | 13 | 3 | 5
Cardiac and Hemodynamic (General) (Cardiac disorders) | 17 | 3 | 7
GI (General) (Gastrointestinal disorders) | 6 | 2 | 2
Arterial (Vascular disorders) | 18 | 7 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acute (N=50) | Sub-acute (N=24) | Chronic (N=26)
Renal Complications (General) (Renal and urinary disorders) | 3 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less